CLINICAL TRIAL: NCT01838213
Title: Extended Spectrum Beta-lactamases - Treatment, Carriage, Environmental Dissemination And Population Epidemiology
Brief Title: Extended Spectrum Betalactamase Producing Bacteria; Epidemiology and Treatment in Non-hospitalized Patients
Acronym: ESCAPE
Status: Completed | Type: Observational
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: Helse Sor-Ost (Other Government); University Hospital of North Norway (Other); University of Oslo (Other)
Responsible Party: Sponsor
Other Study IDs: REK S-08901b
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Results first posted 2015-11-23 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-10

CONDITIONS: Urinary Tract Infection; Infection Due to ESBL Bacteria; Environmental Contamination of ESBL
Keywords: Urinary tract infection; ESBL; treatment; carriage; risk factors; water contamination
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bacterial cultures
Oversight: Data Monitoring Committee: No

SUMMARY:
This project aims at investigating the duration of human fecal carriage of bacteria harboring plasmid-borne resistance genes expressing Extended Spectrum beta-lactamases (ESBL), risk factors for infections with such bacteria and persistence, mobility and spread of ESBL in the environment and within households. It also aims to compare different methods of detecting ESBL carriage and treat patients with urinary tract infection caused by these bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients >=18 of age with a urine culture yielding E. coli or K. pneumoniae >10.000 colony forming units/mL.

Exclusion Criteria:

* Patients who have lived in Norway for <1 year
* Patients who are unable to answer a questionaire
* Patients who have been infected with an ESBL producing bacteria before
* Patients who have been admitted to a hospital or a long term care facility for >24 hours during the past 31 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients living in Eastern Norway who have an urine submitted for culturing to the Department of Medical Microbiology, Vestre Viken Hospital Trust, which covers an area of about 450.000 inhabitants.
  All patients with an bacteria producing ESBL were eligible while patients without ESBL producing bacteria were randomly sampled.
Sampling Method: Non-Probability Sample
Enrollment: 760 (Actual)
Dates: Start 2009-02; Primary Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pål A Jenum, PhD, Study Director — Vestre Viken Hospital Trust

REFERENCES:
- [Result] Soraas A, Sundsfjord A, Jorgensen SB, Liestol K, Jenum PA. High rate of per oral mecillinam treatment failure in community-acquired urinary tract infections caused by ESBL-producing Escherichia coli. PLoS One. 2014 Jan 15;9(1):e85889. doi: 10.1371/journal.pone.0085889. eCollection 2014. PMID 24454943
- [Result] Soraas A, Sundsfjord A, Sandven I, Brunborg C, Jenum PA. Risk factors for community-acquired urinary tract infections caused by ESBL-producing enterobacteriaceae--a case-control study in a low prevalence country. PLoS One. 2013 Jul 23;8(7):e69581. doi: 10.1371/journal.pone.0069581. Print 2013. PMID 23936052
- [Result] Soraas A, Olsen I, Sundsfjord A, Handal T, Bjorang O, Jenum PA. Extended-spectrum beta-lactamase-producing bacteria are not detected in supragingival plaque samples from human fecal carriers of ESBL-producing Enterobacteriaceae. J Oral Microbiol. 2014 Aug 20;6. doi: 10.3402/jom.v6.24026. eCollection 2014. PMID 25206941

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with any type of CA-UTI caused by ESBL-producing or non-ESBL producing E. coli and receiving empirical treatment were included in the study. Data on treatment outcome were obtained and possible associations between outcome and mecillinam treatment, ESBL-status and other variables were investigated.
Groups:
- Patients With UTI Caused by Extended-spectrum β-lactamase-prod: Patients with UTI caused by extended-spectrum β-lactamase-producing E. coli
- Patients With UTI Caused by Non-ESBL-producing E. Coli: Patients with UTI caused by non-ESBL-producing E. coli
Period: Overall Study
Arm/Group | Patients With UTI Caused by Extended-spectrum β-lactamase-prod | Patients With UTI Caused by Non-ESBL-producing E. Coli
Started | 247 | 453
Completed | 81 | 262
Not Completed | 166 | 191
Not completed — Ineligible | 166 | 191

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients With UTI Caused by Extended-spectrum β-lactamase-prod | Patients With UTI Caused by Non-ESBL-producing E. Coli | Total
Number analyzed (Participants) | 81 | 262 | 343
Age, Continuous [Mean (Full Range); unit: years] | 54 [18 to 92] | 61 [19 to 93] | 59 [18 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 225 | 300
  Male | 6 | 37 | 43
Region of Enrollment [Number; unit: participants]
  Norway | 81 | 262 | 343

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failure
Description: Patients included in the study with urinary tract infection (UTI) and treated as part of normal routine were followed for 14 days and further prescriptions of antimicrobials normally used for treatment of UTI will be considered treatment failures. Only participants that received pivmecillinam are reported here. In the paper published in PlosOne "High Rate of Per Oral Mecillinam Treatment Failure in Community-Acquired Urinary Tract Infections Caused by ESBL-Producing Escherichia coli" the mecillinam treatment group were compared with the group that did not receive mecillinam.
Time Frame: 14 days after initiation of treatment
Population: Patients that did receice pivmecillinam.
Measure: Number; unit: Treatment success
Arm/Group | Patients With UTI Caused by Extended-spectrum β-lactamase-prod | Patients With UTI Caused by Non-ESBL-producing E. Coli
Number analyzed (Participants) | 41 | 117
Treatment success | 23 | 101

2. Secondary Outcome: Subjective Outcome
Description: A patient form will be filled in. Data about cessation of symptoms of urinary tract infection will be recorded.
Time Frame: 14 days
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Carriage of ESBL Producing Bacteria
Description: Culture results from patient fecal samples will be collected up to 3 years after urinary tract infection and carriage of ESBL producing bacteria will be examined.
Time Frame: up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Participants in the study were treated for their urinary tract infection as part of routine and adverse events were not recorded.
Arm/Group | Patients With UTI Caused by Extended-spectrum β-lactamase-prod | Patients With UTI Caused by Non-ESBL-producing E. Coli
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/262
Other Adverse Events (participants affected / at risk) | 0/81 | 0/262

LIMITATIONS AND CAVEATS:
Publication of results:

"High Rate of Per Oral Mecillinam Treatment Failure in Community-Acquired Urinary Tract Infections Caused by ESBL-Producing Escherichia coli http://journals.plos.org/plosone/article?id=10.1371/journal.pone.0085889

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes